CLINICAL TRIAL: NCT05879601
Title: "Comparative Evaluation of 3 Dimensional Changes of Dentition in Post Orthodontic Patients With Immediate vs Delayed (Post 24 Hours) Retainer Delivery-A Randomized Control Trial"
Brief Title: "Comparative Evaluation of 3 Dimensional Changes of Dentition in Post Orthodontic Patients With Immediate vs Delayed (Post 24 Hours) Retainer Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PGIDS/BHRC/22/33 Sidhant Goyal
Record Dates: First submitted 2022-07-27; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Relapse
Keywords: Orthodontic Retention
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group- immediate retainer delivery (Other): Retainer will be given to the patients immediately [ Just after debonding]
  Interventions: Other: immediate orthodontic retainer delivery
- experimental group- delayed retainer delivery (Active Comparator): Retainer will be given to the patient 24 hours post debonding.
  Interventions: Other: delayed orthodontic retainer delivery.

INTERVENTIONS:
Other: immediate orthodontic retainer delivery — post orthodontic treatment patients will be given orthodontic retainer immediately after debonding.
  Arms: control group- immediate retainer delivery
Other: delayed orthodontic retainer delivery. — post orthodontic treatment patients will be given orthodontic retainer after 24 hours of debonding.
  Arms: experimental group- delayed retainer delivery

SUMMARY:
Orthodontic treatment goals can be expressed as achieving ideal tooth alignment, esthetic, functional occlusion and stability. Various occlusal changes occur after active phase of orthodontic treatment, these unwanted changes are called relapse. Reitan pointed out that major percentage of changes following active phase of treatment is seen within 24 hours.

To alleviate the effect of relapse, retention is needed. There is little agreement among clinicians about orthodontic retention protocol due to insufficient evidence in the literature on 1. time of retainer delivery 2. unexpected post- treatment changes. 3.quantification of relapse tendency.

The present study will be undertaken to assess the changes and compare if there is any difference in the movement of teeth in post orthodontic treatment cases with immediate and delayed (post 24 hours) retainer delivery.

Thus help in deciding when should the retainer delivery is preffered.

DETAILED DESCRIPTION:
The proposed study will be a prospective, non-pharmacological, single blind, randomized clinical trial to evaluate if there is a difference in transverse (Xaxis), A-P(Y-axis) and Vertical plane(Z-axis) of dentition in two group of post orthodontic treatment patients with immediate retainer delivery in one group and post 24 hours retainer delivery in other group of patients. The present study will be conducted in the Department of Orthodontic and Dentofacial Orthopedics, P.G.I.D.S, Pt. B.D Sharma University of health sciences, Rohtak. The study will be carried out after the institutional approval obtained from ethical committee.

A sample size of 18 patients was calculated keeping confidence interval 95% with power 80%. Accounting for a 10% drop out rate, 20 patients will be enrolled in each group. Patient will be randomly allocated to the study group by a person not involved in the trial using computer generated randomization list. Changes in the tooth movement in transverse(X-axis), A-P(Y-axis), Vertical plane(Zaxis) will be compared in terms of intercanine width, intermolar width, overjet, overbite and contact point displacement between the two groups at following time intervals. These parameters will be charted at T0, T1, T2,T3 and T4 for each patient.Changes in the tooth movement in transverse(X-axis), A-P(Y-axis), Vertical plane(Z-axis) will be compared in terms of intercanine width, intermolar width, overjet, overbite and contact point displacement between the two groups at following time intervals. These parameters will be charted at T0, T1, T2,T3 and T4 for each patient. T0 - Baseline records, at the time of debonding. T1 - Records obtained at the time of retainer delivery. T2 - Records obtained after 1 month of retainer delivery. T3 - Records obtained after 3 months of retainer delivery. T4 - Records obtained after 6 months of retainer delivery

ELIGIBILITY:
Inclusion Criteria:

* Adult orthodontic patients treated with 022*028 MBT appliance with following sequence of wires- 014, 016, 16*22, 17*25, 19*25 NiTi followed by 19*25 SS.
* Treatment duration of 24-36 months with Optimal functional occlusion at end of treatment (PAR score >70%).
* Class I bimax and Class II div I with pre-treatment Little's irregularity index <6mm in both upper and lower arch.
* Nonsurgical and non-orthopedic patients.
* Non syndromic patients and no impaction of teeth except third molars.
* No previous orthodontic treatment.
* Optimal periodontal condition and Good oral hygiene.
* Good compliance regarding retainer wear (Cases who never missed more than 2 consecutive appointment and who reported with less no of breakages)

Exclusion Criteria:

* Subjects with incomplete orthodontic treatment.
* TMJ disorder patients.
* Any systemic disease affecting bone and general growth.
* Patients with incomplete records.
* Patient who fail to follow up or undergo complete treatment.
* Patient with learning difficulties

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-12-25 (Estimated); Study Completion 2024-04-25 (Estimated)

PRIMARY OUTCOMES:
Overjet | T0 - baseline on the day of debonding
  sagittal distance between upper and lower incisors
Overjet | T1 - 24 hours after debonding
  sagittal distance between upper and lower incisors
Overjet | T2 - 1 month after debonding
  sagittal distance between upper and lower incisors
Overjet | T3 - 3 month after debonding
  sagittal distance between upper and lower incisors
Overjet | T4 - 6 month after debonding
  sagittal distance between upper and lower incisors
contact point displacement | T0 - baseline on the day of debonding
  displacement of contact points in anterior teeth
contact point displacement | T1 - 24 hours after debonding
  displacement of contact points in anterior teeth
contact point displacement | T2 - 1 month after debonding
  displacement of contact points in anterior teeth
contact point displacement | T3 - 3 month after debonding
  displacement of contact points in anterior teeth
contact point displacement | T4 - 6 month after debonding
  displacement of contact points in anterior teeth
overbite | T0 - baseline on the day of debonding
  vertical overlap of upper and lower incisors
overbite | T1 - 24 hours after debonding
  vertical overlap of upper and lower incisors
overbite | T2 - 1 month after debonding
  vertical overlap of upper and lower incisors
overbite | T3 - 3 month after debonding
  vertical overlap of upper and lower incisors
overbite | T4 - 6 month after debonding
  vertical overlap of upper and lower incisors
intermolar width | T0 - baseline on the day of debonding
  transverse distance between the first molars
intermolar width | T1 - 24 hours after debonding
  transverse distance between the first molars
intermolar width | T2 - 1 month after debonding
  transverse distance between the first molars
intermolar width | T3 - 3 month after debonding
  transverse distance between the first molars
intermolar width | T4 - 6 month after debonding
  transverse distance between the first molars
intercanine width | T0 - baseline on the day of debonding
  transverse distance between the canine
intercanine width | T1 - 24 hours after debonding
  transverse distance between the canine
intercanine width | T2 - 1 month after debonding
  transverse distance between the canine
intercanine width | T3 - 3 month after debonding
  transverse distance between the canine
intercanine width | T4 - 6 month after debonding
  transverse distance between the canine

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No